CLINICAL TRIAL: NCT00243178
Title: A Parallel Randomized Controlled Evaluation of Clopidogrel Plus Aspirin, With Factorial Evaluation of Irbesartan, for the Prevention of Vascular Events, in Patients With Atrial Fibrillation
Brief Title: Atrial Fibrillation Clopidogrel Trial With Irbesartan for Prevention of Vascular Events (ACTIVE W)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: ICD Study Director, Sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EFC4912 W
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Atrial Fibrillation; Vascular Risk
Keywords: Atrial fibrillation; Anticoagulant therapy; Thromboembolic prevention
MeSH Terms: conditions — Atrial Fibrillation | interventions — Clopidogrel

INTERVENTIONS:
Drug: clopidogrel (SR25990C) — 75 mg once daily in combination with aspirin

SUMMARY:
The purpose of this study is to determine if the combination of Clopidogrel 75mg once daily (od) plus aspirin at 100mg daily (recommended dose) is as effective as oral anticoagulation therapy with a lower risk of bleeding in patients with atrial fibrillation associated with at least one major cardiovascular risk factor.Primary objectives :The combination of clopidogrel plus aspirin compared to adjusted dose (INR between 2.0 and 3.3) oral anticoagulation (a vitamin K antagonist) will result in the same risk of the composite outcome of stroke, non-CNS systemic embolism, myocardial infarction or vascular death in patients with atrial fibrillation.The secondary objective is to establish whether or not aspirin plus clopidogrel has a lower risk of hemorrhage than standard anticoagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of atrial fibrillation either on one current Electrocardiogram (ECG) or on two ECG recorded at two weeks a part during 6 months prior to study enrollment.
* Evidence of high risk of vascular events: at least one of the following risk criteria must be present:

  * are 75 years or greater;
  * on treatment for systemic hypertension;
  * prior stroke, TIA, or non-CNS systemic embolus;
  * left ventricular dysfunction with left ventricular ejection fraction (EF) estimated by echocardiogram or angiogram (radionuclide or contrast) to be < 45%;
  * peripheral vascular disease (previous peripheral artery revascularization, limb and foot amputation, or the combination of current intermittent claudication and ankle arm systolic blood pressure ratio < 0.9);
  * age 55 to 74 years; AND
  * either diabetes mellitus requiring drug therapy, or documented previous myocardial infarction, or documented coronary artery disease.

Exclusion Criteria:

* Patients will be excluded from ACTIVE if any of the following are present :

  * requirement for clopidogrel (such as recent coronary stent procedure);
  * requirement for oral anticoagulant (such as prosthetic mechanical heart valve);
  * prior intolerance to ASA or clopidogrel;
  * documented peptic ulcer disease within the previous 6 months;
  * prior intracerebral hemorrhage;
  * significant thrombocytopenia; (platelet count < 50 x 10(9)/L);
  * psychosocial reason making study participation impractical;
  * geographic reason making study participation impractical;
  * ongoing alcohol abuse;
  * mitral stenosis;
  * pregnant or nursing woman or woman of child bearing potential and not on effective birth control for at least one month prior to start of study or not willing to continue on birth control for duration of study;
  * severe comorbid condition such that the patient is not expected to survive 6 months;
  * patient currently receiving an investigational pharmacologic agent; OR
  * requirement for chronic (> 3 months) non-COX-2 inhibitor NSAID therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6706 (Actual)
Dates: Start 2003-07; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome:time to the first occurrence of stroke, non-CNS systemic embolism, myocardial infarction or vascular death | during approximately three years of follow-up

SECONDARY OUTCOMES:
Secondary outcomes: major hemorrhage, total mortality and stroke. | during approximately three years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Salim YUSUF, Prof., Study Chair — Hamilton Health Sciences Corporation
Locations (32):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Result] ACTIVE Writing Group of the ACTIVE Investigators; Connolly S, Pogue J, Hart R, Pfeffer M, Hohnloser S, Chrolavicius S, Pfeffer M, Hohnloser S, Yusuf S. Clopidogrel plus aspirin versus oral anticoagulation for atrial fibrillation in the Atrial fibrillation Clopidogrel Trial with Irbesartan for prevention of Vascular Events (ACTIVE W): a randomised controlled trial. Lancet. 2006 Jun 10;367(9526):1903-12. doi: 10.1016/S0140-6736(06)68845-4. PMID 16765759
- [Derived] Flaker GC, Pogue J, Yusuf S, Pfeffer MA, Goldhaber SZ, Granger CB, Anand IS, Hart R, Connolly SJ; Atrial Fibrillation Clopidogrel Trial With Irbesartan for Prevention of Vascular Events (ACTIVE) Investigators. Cognitive function and anticoagulation control in patients with atrial fibrillation. Circ Cardiovasc Qual Outcomes. 2010 May;3(3):277-83. doi: 10.1161/CIRCOUTCOMES.109.884171. Epub 2010 Mar 16. PMID 20233976
- [Derived] Cairns JA, Wittes J, Wyse DG, Pogue J, Gent M, Hirsh J, Marler J, Pritchett EL. Monitoring the ACTIVE-W trial: some issues in monitoring a noninferiority trial. Am Heart J. 2008 Jan;155(1):33-41. doi: 10.1016/j.ahj.2007.09.011. Epub 2007 Nov 26. PMID 18082486
- [Derived] Hohnloser SH, Pajitnev D, Pogue J, Healey JS, Pfeffer MA, Yusuf S, Connolly SJ; ACTIVE W Investigators. Incidence of stroke in paroxysmal versus sustained atrial fibrillation in patients taking oral anticoagulation or combined antiplatelet therapy: an ACTIVE W Substudy. J Am Coll Cardiol. 2007 Nov 27;50(22):2156-61. doi: 10.1016/j.jacc.2007.07.076. Epub 2007 Nov 13. PMID 18036454